CLINICAL TRIAL: NCT03568526
Title: The Effects of a Sensorimotor Rehabilitation Program on the Upper and Lower Limbs of Persons With Cancer Following Taxane-Based Chemotherapy for Early Stage Breast Cancer
Brief Title: Sensorimotor Rehabilitation Program in Improving Quality of Life in Patients With Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Amy Darragh, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-14219; NCI-2017-01583 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-03-20; First posted 2018-06-26 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Peripheral Neuropathy; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (sensorimotor rehabilitation program) (Experimental): Patients attend 1 therapy session to receive education and training in the use of the home program. Patients then complete exercises over 90 minutes per week for 6 weeks.
  Interventions: Other: Educational Intervention; Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Attend a therapy session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Exercise Intervention — Complete exercise
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well the sensorimotor rehabilitation program works in improving quality of life in patients with early stage breast cancer. A hand and foot sensory improvement program from occupational and physical therapists may improve patients' function in everyday tasks and overall quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the effects of an innovative, new sensorimotor rehabilitation program on persons with cancer following taxane-based chemotherapy for early stage breast cancer.

OUTLINE:

Patients attend 1 therapy session to receive education and training in the use of the home program. Patients then complete exercises over 90 minutes per week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a primary diagnosis of grade 1 or greater peripheral neuropathy of the upper and lower extremities
* Taxane-based chemotherapy for early stage breast cancer
* Diagnosis of early stage breast cancer

Exclusion Criteria:

* Individuals with late stage breast cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Identify differences in patients scores using post-test scores on the McGill Pain Questionnaire | Up to 2 years
  The McGill Pain Questionnaire-Short Form (MPQ-SF). The purpose of the MPQ-SF is to rate qualities and intensities of pain. Fifteen words describe pain and the subject rates the pain words using a 4-point Likert scale. A visual analogue scale is used to identify intensity of pain and symptoms are rated on current and length of pain. The MPQ-SF has been shown to be a valid and reliable tool in the assessment of pain and specifically the assessment of cancer pain.7.8,9 The Breast Edge Task Force Outcomes Committee rated the MPQ-SF as "highly recommend" for use in the breast cancer population.
Evaluate patients using post-test scores on the CIPN-20 | Up to 2 years
  The purpose of the CIPN-20 is to identify quality of life. Twenty items are used to identify symptoms and functional limitations related to CIPN. Three subscales represent sensory, motor, and autonomic function and provide a more complete picture of the nature, frequency, and severity of CIPN. The CIPN-20 is a multidimensional scale that was specifically developed to capture patients' symptoms and functional limitations as related to CIPN 11,12. The CIPN-20 is best utilized when combined with other pain and quality of life tools.
Assess the differences in patients post-test scores on the Disability of Arm Hand and Shoulder scores | Up to 2 years
  The purpose of the Quick-DASH is to measure physical function and symptoms of persons with musculoskeletal disorders of the upper limb. 3 It is a shortened version of the DASH, using 11 items instead of 30. In the breast cancer population, the DASH has shown good outcome measures when testing physical, social and psychological concerns.13,14 The DASH is highly recommended in the breast cancer population and the Quick DASH is also recommended but has not been used as frequently in research.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Darragh, PhD, OTR/L, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu